CLINICAL TRIAL: NCT04433078
Title: RepurpoSing Old Drugs TO SuppRess a Modern Threat: The STORM Trial
Brief Title: RepurpoSing Old Drugs TO SuppRess a Modern Threat: COVID-19 STORM
Acronym: STORM
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No Participants Enrolled
Sponsor: Temple University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: The STORM Trial
Record Dates: First submitted 2020-06-10; First posted 2020-06-16 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Cytokine Storm; SARS-CoV-2
Keywords: Doxycycline; Cytokine Storm; SARS-CoV-2
MeSH Terms: conditions — Cytokine Release Syndrome | interventions — Doxycycline

STUDY DESIGN:
Intervention Model Description: This study will randomize 20 patients with confirmed or highly suspected early stage severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) patients to Doxycycline (100 mg BID) or Placebo.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Doxycycline (Experimental): Participants receive 100 MG BID for 21 days
  Interventions: Drug: Doxycycline
- Placebo (Placebo Comparator): Participants receive Placebo BID for 21 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Doxycycline — 100 MG Tablet
  Arms: Doxycycline
Drug: Placebo — Placebo Tablet
  Arms: Placebo

SUMMARY:
The primary aim of this study is to test whether Doxycycline can benefit patients with severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infections by inhibiting the replication of the virus while at the same time blocking the development of cytokine storms or inhibiting cytokine-associated coagulopathy respectively. The investigators hypothesize that Doxycycline will will improve survival and reduce morbidity in SARS-CoV-2 infected patients.

A secondary aim is to identify genetic variants that predict either an unusually mild disease or an unusually severe disease - knowledge that can be used to design new and precise medications and to be able to predict patients who might get into early trouble and to therefore hospitalize them.

DETAILED DESCRIPTION:
This study will randomize 20 patients with confirmed or highly suspected early stage severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) to Doxycycline (100 mg BID) or Placebo and then assess the progression of their disease over the next three weeks with the primary endpoint being days alive and out of the hospital.

The investigators will collect specimens for measurement of viral burden (nasopharyngeal luminex (SARS-CoV-2), SARS-CoV-2 serum quantitative viral load, SARS-CoV-2 IgM/IgG antibodies), markers of inflammation (WBC, ESR, TNFa, IL-1, IL-6, IL-1B), and cardiac dysfunction (CRP, pro-BNP, hsTnT).

Eligibility will be based on history and physical examination findings - collated into a clinical suspicion score. The decision to enroll based on clinical suspicion score rather than confirmed SARS-CoV-2 disease is based on the variable and unacceptably high false negative rate of the nasopharyngeal PCR test for in early disease.

Clinical Suspicion Score: Greater than or equal to 6/20 (at least 4 points of which must be clinical) will be eligible for enrollment.

Clinical Criteria: Max 12 points

* Fever (2 points)
* Cough (2 points)
* Dyspnea (2 points)
* Chest pain (1 point)
* Myalgias (1 point)
* Fatigue (1 point)
* GI symptoms (1 point)
* Loss of Smell (1 point)
* Loss of Taste (1 point)

Exposure Criteria: Max 8 points

* Contact with known COVID+ (2 points)
* Healthcare worker -- frequent <6 feet contact for 15 minutes (2 points)
* High-risk work -- supermarket, deli, transportation (2 points)
* Endemic community -- prison/jail/nursing home/LTAC/SNF/rehab/homeless/homeless shelter (2 points)

Genetic variants may explain why patients who are infected with SARS-CoV-2 have either a relatively benign or an inappropriately aggressive response to an infectious insult. Medications may be more or less effective in that group of patients harboring genetic variants of a disease-related protein. To better understand this, whole genome sequencing and analysis will be performed on all study patients.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed or highly suspected early stage severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), disease with clinical suspicion score >6/20, not requiring hospitalization
* Age ≥18 years
* Willing to sign the informed consent form
* Willing to take study drug or placebo as directed for 21 days

Exclusion Criteria:

* Confirmed or highly suspected early stage severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), disease with clinical suspicion score >6/20, requiring hospitalization
* Suspected or confirmed convalescent severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), within the prior 4 weeks
* Age <18 years' old
* Inability to take medications orally
* Inability to provide written consent
* Known sensitivity/allergy to doxycycline or tetracyclines
* Current use of doxycycline for another indication
* Pregnancy
* A known diagnosis of myasthenia gravis
* History of Clostridium Difficile infection within past 12 months
* Sun sensitivity
* Individuals using medications which could lower doxycycline levels, including barbiturates, phenytoin, carbamazepine, warfarin
* Individuals using isotretinoin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06-22 (Actual); Primary Completion 2021-04-13 (Actual); Study Completion 2021-04-13 (Actual)

PRIMARY OUTCOMES:
Time Free of Either Hospitalization, Hypoxemia, ICU Admission or Death | 21 days
  Days Alive and Out of Hospital (Composite Endpoint)

SECONDARY OUTCOMES:
NP SARS-CoV-2 PCR | 21 days
  Change From Baseline of Nasopharyngeal Luminex NxTAG CoV (Positive/Negative)
SARS-CoV-2 Serum Quantitative Viral Load | 21 days
  Change From Baseline of SARS-CoV-2 Serum Quantitative Viral Load
SARS-CoV-2 IgM/IgG Antibodies | 21 days
  Change From Baseline of SARS-CoV-2 IgM/IgG Antibodies (Positive/Negative)
White Blood Cell Count (WBC) | 21 days
  Change From Baseline of White Blood Count (CBC) K/mm3
Absolute Lymphocyte Count (ALC) | 21 days
  Change From Baseline of Absolute Lymphocyte Count (ALC) K/mm3
C-Reactive Protein (CRP) | 21 days
  Change From Baseline of C-Reactive Protein (CRP) mg/dL
N-Terminal Pro-B-Type Natriuretic Peptide (Pro-BNP) | 21 days
  Change From Baseline of N-Terminal Pro-B-Type Natriuretic Peptide (Pro-BNP) pg/mL
High Sensitivity Troponin I (hsTnT) | 21 days
  Change From Baseline of High Sensitivity Troponin I (hsTnT) ng/mL
Tumor Necrosis Factor Alpha (TNF-a) | 21 days
  Change From Baseline of Tumor Necrosis Factor Alpha (TNF-a)
IL-1 | 21 days
  Change From Baseline of IL-1
IL-1B | 21 days
  Change From Baseline of IL-1B
IL-6 | 21 days
  Change From Baseline of IL-6

CONTACTS AND LOCATIONS:
Overall Officials: Arthur M Feldman, MD, PhD, Principal Investigator — Temple University
Locations (1):
- Temple University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No